CLINICAL TRIAL: NCT04283617
Title: Reversibility of Brain Glucose Transport and Metabolism in T2DM: an Intervention Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to funding issues.
Sponsor: Yale University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000027293; 1KL2TR001862-01 (NIH)
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Diabete Type 2
Keywords: continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nutritional Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic with short duration (Experimental): Type 2 diabetics with HbA1c > 7.5 % with short duration of diabetes < 5 years
  Interventions: Behavioral: Intensification of insulin regimen/Nutrition
- Diabetic with long duration (Experimental): Type 2 diabetics with HbA1c > 7.5 % with short duration of diabetes > 5 years
  Interventions: Behavioral: Intensification of insulin regimen/Nutrition

INTERVENTIONS:
Behavioral: Intensification of insulin regimen/Nutrition — The intensification of the diabetes regimens will be managed by Dr. Sanchez Rangel, a fully trained attending endocrinologist, The weight goal will be to have no more than 5% weight change. Participants will have regular phone and in-person MD and nutritionist communication over the course of the 12-week study. All individuals will be asked to perform SMBG at least 4 times a day (before breakfast, lunch, dinner, and bedtime). The daily SMBG records will be sent to Dr. Sanchez Rangel weekly for review to guide adjustment of insulin regimens. Target blood glucose levels will be between 80-130 mg/dl before meals and between < 180 mg/dl at bedtime. Throughout the study, individuals will be contacted via telephone call, email or through additional clinic visits as deemed necessary for maintenance of glycemic control. All individuals will receive education regarding the detection and proper management of hypoglycemia.

SUMMARY:
This study is designed to test if there is a difference in brain glucose transport kinetics in poorly controlled T2DM individuals with short duration and long duration of diabetes, using non-invasive magnetic resonance spectroscopy (MRSI). Also, if these changes are reversible with improved glucose control will be tested. A better understanding of the impact of duration of diabetes on brain glucose transport function may have important implications for understanding the pathophysiology of brain complications in T2DM.

DETAILED DESCRIPTION:
Specific Aim 1: To compare brain glucose transport and metabolism in age, BMI, and HbA1c matched T2DM individuals with either long duration of diabetes or short duration of diabetes using brain 1H MRSI during hyperglycemic clamp

Hypothesis: T2DM individuals with chronic uncontrolled diabetes will have lower brain glucose levels as compared with age, BMI, and HbA1c matched T2DM individuals with shorter duration of diabetes.

Screening visit: Volunteers will be screened at the Yale New Haven Hospital (YNHH) Hospital Research Unit (HRU) or Yale Center for Clinical Investigation (YCCI) Church street Research Unit (CSRU) with a medical history and exam. Blood tests will be collected for A1C, ALT, TSH, Hgb and Creatinine. A urine pregnancy test will be performed on all women of childbearing potential, and women who are pregnant will be excluded.

Continuous Glucose Monitoring (CGM): Participants will wear for 14 days prior to the MRSI scanning sessions a CGM (FreeStyle Libre Pro glucose monitoring system) to continuously monitor their interstitial blood glucose levels. Given that this data is blinded, patients will be informed that it is not a replacement for self-monitoring of blood glucose. Subjects should continue their normal testing routine while wearing the sensor. CGM placement will take place at the HRU or CSRU. Those not already using CGM in their usual care will be trained in its proper use by experienced study staff. Patients already using CGM will be allowed to use their usual CGM, however, they will also be asked to wear a second blinded study sensor. Subjects will be provided with our contact information in the event that they have any questions, concerns or issues related to the CGM. Intense exercise may cause the sensor to loosen due to sweat or movement of the sensor. If the CGM sensor falls off while the subject is wearing it, subjects will be asked to return to the HRU or CSRU so that a new sensor can be re-inserted.

The CGM consists of a sensor that measures glucose levels from the interstitial tissue. The sensor is sterile and comes in an unopened package. It has a plastic wire-like tip that is placed under the skin and continuously measures the glucose levels. A trained study staff member will insert the CGM wirelike tip under the volunteer's skin with the use of the CGM sensor insertion kit. Each sensor is single use only and disposable. The FreeStyle Libre Pro does not require any calibration, as is the case with other CGM devices. This means that no finger sticks are required for its use.

CGM removal: After 14 days of wearing the CGM, it will be removed by a trained study staff member on the on the same day as the subject's scan. To remove the sensor, the adhesive patch will be gently peeled off from the skin, together with the sensor. Removal of the sensor is a painless procedure. The sensor will be discarded after use.

MRSI scanning and Hyperglycemic Clamp: Participants will arrive at MRRC at 7AM on the morning of the study after an 8 hour overnight fast. A urine pregnancy test will be performed on all women of childbearing potential, and women who are pregnant will be excluded. Following IV placements and baseline blood collection, at ~8 AM all T2DM subjects will receive insulin infusion to keep plasma glucose levels at ~100-110 mg/dl. Once glucose levels are stabilized, the subjects will be transferred into the 4T scanner for the hyperglycemia clamp.

Subjects will lie supine in a 4.0 T whole-body magnet interfaced to a Bruker AVANCE spectrometer (Bruker Instruments) with the head immobilized with foam inserts on top of a radiofrequency probe consisting of a 1H coil, as previously described by our group. A nurse experienced with working in a MRS environment will be with subjects at all times. If patients express discomfort or anxiety and ask to be removed from the scanner, the session will be immediately terminated.

Following the 45-minute baseline scan, subjects will remain in the scanner for continuous scanning during the hyperglycemic clamp. An infusion of 20% dextrose at a variable rate to maintain plasma glucose levels at 220 mg/dL for 2 hours. Glucose infusion rates will be adjusted in response to plasma glucose levels measured every 5-10 minutes. Subjects will be able to take breaks as needed during the 2 hours hyperglycemic clamp and MRS scan. During the clamp study a series of hormones will be obtained including insulin levels, GLP1, leptin and free fatty acids.

Neurocognitive testing: Participants will undergo a panel of cognitive testing to assess working memory, learning and executive function; visual, verbal and episodic memory; attention, information processing and reaction time; social and emotion recognition, decision making and response control (CANTAB Cognitive research software, Cambridge Cognition).

Specific Aim 2: To assess the impact that duration of diabetes has on reversibility of brain glucose transport kinetics as assessed by 1H MRSI scanning before and after a 12-week intervention to improve glycemic control

Hypothesis: Participants with shorter duration of diabetes (<5 years) will have greater magnitude of restoration of brain glucose transport parameters compared to T2DM participants with longer duration of diabetes (>5 years).

Subjects: Subjects from Aim 1 will undergo intensification of their diabetes management for a period of 12-week and at the end of the intervention they will undergo 1H MRSI scanning to measure intracerebral and plasma glucose levels at euglycemia and following 2 hours of hyperglycemia using the clamp technique (target glucose 220 mg/dl) in the occipital region. (Figure 2)

Intensification of insulin regimen/Nutrition visit:

The intensification of the diabetes regimens will be managed by Dr. Sanchez Rangel, a fully trained attending endocrinologist, and will follow the general strategies outlined in the Position Statement of the American Diabetes Association and the European Association for the Study of Diabetes. All participants will receive exercise and dietary counseling from Mary Savoye, a nutritionist and registered dietician with extensive experience with working with individuals with diabetes and obesity, and who has worked with Dr. Sanchez Rangel on her current pilot. The weight goal will be to have no more than 5% weight change. Participants will have regular phone and in-person MD and nutritionist communication over the course of the 12-week study. All individuals will be asked to perform SMBG at least 4 times a day (before breakfast, lunch, dinner, and bedtime). The daily SMBG records will be sent to Dr. Sanchez Rangel weekly for review to guide adjustment of insulin regimens. Target blood glucose levels will be between 80-130 mg/dl before meals and between < 180 mg/dl at bedtime. Individuals not at goal glycemic targets will undergo intensification of their regimen. Throughout the study, individuals will be contacted via telephone call, email or through additional clinic visits as deemed necessary for maintenance of glycemic control. All individuals will receive education regarding the detection and proper management of hypoglycemia.

Continuous Glucose Monitoring (CGM): Identical to Aim 1.

MRSI scanning and Hyperglycemic Clamp: Study design will be identical to Aim 1

Neurocognitive testing: Study design will be identical to Aim 1

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetics with HbA1c > 7.5% with short duration of diabetes <5 years or
* Type 2 Diabetics with HbA1c > 7.5% longer duration of diabetes >5 years

Exclusion Criteria:

* Patients treated with incretin-based therapies
* Creatinine > 1.5 mg/dL
* Hgb < 10 mg/dL
* ALT > 3 X ULN
* Untreated thyroid disease
* Uncontrolled hypertension
* Known neurological disorders
* Untreated psychiatric disorders
* Malignancy
* Bleeding disorders
* Smoking
* Current or recent steroid use in last 3 months
* Illicit drug use
* Women: pregnancy, actively seeking pregnancy, or breastfeeding
* Inability to enter MRI/MRS (per standard MRI safety guidelines)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Intracerebral concentrations of glucose | Baseline
  Intracerebral concentrations of glucose across multiple brain locations, including frontal and occipital, as measured by MRSI will be compared following hyperglycemic clamp in uncontrolled T2DM individuals with short duration of diabetes and long duration of diabetes
Intracerebral concentrations of glucose between T2DM patients | 12 Weeks
  Intracerebral concentrations of glucose will be compared between T2DM patients before and after 12 weeks of intensification of their diabetes management

SECONDARY OUTCOMES:
Verbal Recognition Memory (VRM) | Baseline
  Verbal Recognition Memory assesses verbal memory and new learning. It measures the ability to encode and subsequently retrieve verbal information, with recall tapping into fronto temporal networks and recognition assessing hippocampal areas. Administration time: 10 minutes
Verbal Recognition Memory (VRM) | 12 Week
  Verbal Recognition Memory assesses verbal memory and new learning. It measures the ability to encode and subsequently retrieve verbal information, with recall tapping into fronto temporal networks and recognition assessing hippocampal areas. Administration time: 10 minutes
Paired Associates Learning (PAL) | Baseline
  Paired Associates Learning assesses visual memory and new learning. Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed. Administration time: 8 minutes
Paired Associates Learning (PAL) | 12 Week
  Paired Associates Learning assesses visual memory and new learning. Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed. Administration time: 8 minutes
Spatial Working Memory (SWM) | Baseline
  Spatial Working Memory requires retention and manipulation of visuospatial information. This self-ordered test has notable executive function demands and provides a measure of strategy as well as working memory errors. Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes which have already been found to contain a token) and strategy and latency. Administration time: 4 minutes
Spatial Working Memory (SWM) | 12 Week
  Spatial Working Memory requires retention and manipulation of visuospatial information. This self-ordered test has notable executive function demands and provides a measure of strategy as well as working memory errors. Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes which have already been found to contain a token) and strategy and latency. Administration time: 4 minutes
Reaction Time (RTI) | Baseline
  Reaction Time provides assessments of motor and mental response speeds, as well as measures of movement time, reaction time, response accuracy and impulsivity. Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants. Administration time: 3 minutes
Reaction Time (RTI) | 12 Week
  Reaction Time provides assessments of motor and mental response speeds, as well as measures of movement time, reaction time, response accuracy and impulsivity. Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants. Administration time: 3 minutes
Pattern Recognition Memory (PRM) | Baseline
  Pattern Recognition Memory is a test of visual pattern recognition memory in a 2-choice forced discrimination paradigm.Outcome measures include the number and percentage of correct trials and latency (speed of participant's response). Administration time: 4 minutes
Pattern Recognition Memory (PRM) | 12 Week
  Pattern Recognition Memory is a test of visual pattern recognition memory in a 2-choice forced discrimination paradigm.Outcome measures include the number and percentage of correct trials and latency (speed of participant's response). Administration time: 4 minutes
Delayed Matching to Sample (DMS) | Baseline
  Delayed Matching to Sample assesses both simultaneous visual matching ability and short-term visual recognition memory, for non-verbalizable patterns. Outcome measures include latency (the participant's speed of response), the number of correct patterns selected and a statistical measure giving the probability of an error after a correct or incorrect response. Administration time: 7 minutes
Delayed Matching to Sample (DMS) | 12 Week
  Delayed Matching to Sample assesses both simultaneous visual matching ability and short-term visual recognition memory, for non-verbalizable patterns. Outcome measures include latency (the participant's speed of response), the number of correct patterns selected and a statistical measure giving the probability of an error after a correct or incorrect response. Administration time: 7 minutes
Rapid Visual Information Processing (RVP) | Baseline
  Rapid Visual Information Processing is a measure of sustained attention. Outcome measures cover latency (speed of response), probability of false alarms and sensitivity. Administration time: 7 minutes
Rapid Visual Information Processing (RVP) | 12 Week
  Rapid Visual Information Processing is a measure of sustained attention. Outcome measures cover latency (speed of response), probability of false alarms and sensitivity. Administration time: 7 minutes
Multitasking Test (MTT) | Baseline
  The Multitasking Test is a test of the participant's ability to manage conflicting information provided by the direction of an arrow and its location on the screen and to ignore task-irrelevant information. Outcome measures for the Multitasking Test include response latencies and error scores that reflect the participant's ability to manage multitasking and the interference of incongruent task-irrelevant information on task performance (i.e. a Stroop-like effect).Administration time: 8 minutes
Multitasking Test (MTT) | 12 Week
  The Multitasking Test is a test of the participant's ability to manage conflicting information provided by the direction of an arrow and its location on the screen and to ignore task-irrelevant information. Outcome measures for the Multitasking Test include response latencies and error scores that reflect the participant's ability to manage multitasking and the interference of incongruent task-irrelevant information on task performance (i.e. a Stroop-like effect).Administration time: 8 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT04283617/ICF_000.pdf